CLINICAL TRIAL: NCT06392191
Title: Effects of Liposomal Bupivacaine Combined With Bupivacaine and Dexamethasone for Rhomboid Intercostal Block on Postoperative Pain Following Video-Assisted Thoracoscopic Surgery: A Non-inferiority, Double-blind, Randomized Trial.
Brief Title: Comparison of Bupivacaine Liposomal vs Bupivacaine Combined With Dexamethasone for Postoperative Pain in VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, professor, Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY-226
Record Dates: First submitted 2024-04-08; First posted 2024-04-30 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Thoracic Surgery
Keywords: Rhombic intercostal nerve block; thoracoscopy; Bupivacaine liposomes
MeSH Terms: interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinding of medical staff and investigators: a study coordinator was developed to keep and distribute the randomisation numbers, an independent nurse anaesthetist prepared the medication for the study according to the randomisation result code, because bupivacaine liposomes are milky and bupivacaine is colourless, we set up an independent medication preparer and nerve block operator, and nerve block operators were not permitted to be associated with anaesthesia procedures and postoperative Patient assessment. The anaesthesiologist and the follow-up physician were unaware of the grouping.
  Patients were blinded: all patients were anaesthetised and the nerve block was performed without the patients touching the drugs. The double blinding continued throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine liposomes group (Other): The nerve block puncture needle was imaged and then entered into the fascial space between the rhomboid and extracostal muscles, and liposomal bupivacaine 93 mg and bupivacaine 25mg diluted to 20 ml were injected into this space.
  Interventions: Procedure: Rhombic intercostal nerve block(Received liposomal bupivacaine 93 mg and bupivacaine 25 mg diluted to 20 ml)
- Standard bupivacaine dexamethasone group (Other): The nerve block puncture needle was imaged and then entered into the fascial space between the rhomboid and external intercostal muscles, and a mixture of: receive standard bupivacaine 105 mg diluted to 20 ml with dexamethasone 5 mg was injected into this space.
  Interventions: Procedure: Rhombic intercostal nerve block(Receive standard bupivacaine 105 mg diluted to 20 ml with dexamethasone 5 mg.)

INTERVENTIONS:
Procedure: Rhombic intercostal nerve block(Received liposomal bupivacaine 93 mg and bupivacaine 25 mg diluted to 20 ml) — The patient was placed in lateral recumbency and placed medial to the medial border of the scapula in the oblique sagittal plane using a line array ultrasound probe to identify ultrasound landmarks, trapezius, obliques, intercostals, pleura, and lungs, The block needle was then entered in-plane at the T5 level, with the margins retracting on insertion, and the nerve block perforating needle was imaged and then inserted into the fascial gap between the trapezius and the external intercostal muscles. Receive liposomal bupivacaine 93 mg and bupivacaine 25 mg diluted to 20ml.
  Arms: Bupivacaine liposomes group
Procedure: Rhombic intercostal nerve block(Receive standard bupivacaine 105 mg diluted to 20 ml with dexamethasone 5 mg.) — The patient was placed in lateral recumbency and placed medial to the medial border of the scapula in the oblique sagittal plane using a line array ultrasound probe to identify ultrasound landmarks, trapezius, obliques, intercostals, pleura, and lungs, The block needle was then entered in-plane at the T5 level, with the margins retracting on insertion, and the nerve block perforating needle was imaged and then inserted into the fascial gap between the trapezius and the external intercostal muscles. A mixture of standard bupivacaine 105 mg diluted to 20 ml with dexamethasone 5 mg was received.
  Arms: Standard bupivacaine dexamethasone group

SUMMARY:
The purpose of this study, is to investigate the effectiveness of ultrasound-guided rhombic intercostal nerve block for postoperative pain control in thoracoscopic pulmonary resection with bupivacaine liposomes versus bupivacaine hydrochloride with dexamethasone to assess whether bupivacaine liposomes will produce analgesia superior to bupivacaine hydrochloride with dexamethasone in terms of analgesia effect and duration of analgesia. This study will also evaluate whether liposomal bupivacaine after nerve block improves the quality of postoperative recovery compared to bupivacaine hydrochloride combined with dexamethasone.

DETAILED DESCRIPTION:
Approved by the Ethics Committee of Jiaxing No. 1 Hospital (approval number: 2024-KY-226). This study was enrolled prior to patient enrollment in the clinical trial. Written informed consent was obtained from all participants. The study is expected to be conducted from April 2024 through December 2025. This study enrolls 90 elective thoracoscopic lung resection surgery(including wedge resection, segmentectomy, or lobectomy) patients between the ages of 18-80 years, ASA Physical Status I and III, who had no allergic reaction to the study drug.

Basic monitoring such as electrocardiogram, pulse oximetry, and noninvasive blood pressure were arranged preoperatively. The bupivacaine liposome group was treated with bupivacaine liposome 93 mg combined with bupivacaine 25 mg, and the standard control group was treated with bupivacaine hydrochloride 105 mg combined with dexamethasone 5 mg, and both groups were perfused with saline 20 ml. ultrasound-guided rhombic intercostal muscle nerve block was performed for a total of 20 ml. postoperative analgesia was provided using patient-controlled intravenous analgesia (PCIA), and according to the patients weight and baseline condition. Upon arrival of postoperative patients to the ward, if the patient reports significant pain, defined as the numeric rating scale (NRS), score greater than 3, the first step is to administer one press of the analgesic pump. If the pain persists, the pain management protocol will be initiated. Cumulative PCIA consumption at different postoperative time intervals (including 0-24 hours, 24-48 hours, and 48-72 hours). Quality of Recovery Score (QoR-15) at 72 hours postoperatively, If NRS at 6 hours to 3 months, and patient satisfaction were recorded.Pain assessments were performed at the following time points: 0 hours postoperatively (upon tracheal extubation and patient awakening), 0.5 hours, 2 hours, 4 hours, 12 hours, 24 hours, 48 hours, and 72 hours. Pain score follow-up by telephone at the third month.

ELIGIBILITY:
Inclusion Criteria:

ASA physical status I-III, aged between 18 and 80 years, scheduled for elective thoracoscopic lung resection surgery under general anesthesia with endotracheal intubation (including wedge resection, segmentectomy, or lobectomy) with one or three incisions, expected duration of surgery less than 4 hours, and body mass index (BMI) between 18 and 30 kg/m².

Exclusion Criteria:

1. trauma or emergency patients;
2. patients classified as New York Heart Association (NYHA) functional class 3-4;
3. unstable coronary artery disease patients;
4. patients with renal system diseases (estimated glomerular filtration rate <30 mL/min/1.73 m²);
5. patients with liver system diseases (alanine aminotransferase or aspartate aminotransferase levels exceeding twice the normal value);
6. patients with coagulation disorders, or those who have not discontinued warfarin or novel anticoagulants (such as rivaroxaban, dabigatran) prior to surgery;
7. individuals with a history of alcohol abuse or substance dependence within the past two months;
8. patients with uncontrolled anxiety, schizophrenia, or other psychiatric disorders;
9. pregnant or planning to become pregnant women;
10. individuals with a history of allergy to local anesthetics or investigational drugs. Additionally, patients who refuse to sign the informed consent form will also be excluded;
11. chronic pain syndromes (defined as reflex sympathetic dystrophy or complex regional pain syndrome);
12. chronic opioid use (longer than 3 months or daily morphine equivalents more than 5 mg/day for 1 month).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Area under the curve | 0-48 hours after surgery
  Area under the curve of the numeric rating scale (NRS) scores at rest

SECONDARY OUTCOMES:
Change in functional pain using Brief Pain Inventory (BPI) | Preoperative day one, 6 weeks after surgery, 3 months after surgery
  Compare functional pain using the BPI at baseline, 6 weeks and 3 months. The BPI scale defines pain as follows: Score: 1 - 4 = Mild Pain, Score: 5 - 6 = Moderate Pain, Score: 7 - 10 = Severe Pain.
Change in Quality of Recovery 15 questionnaire | Preoperative day one；Day 1, 2 and 7 after surgery
  15 questions assessing the quality of recovery, rated on a ten-point scale with a total score ranging from 0 (very poor recovery) to 150 (good recovery)
Change in white blood cell count (WBC) | Preoperative day one, day 0, day 1 and day 2 after surgery
  Compare the change in postoperative WBC from baseline only for participants that have an overnight hospital stay
Length of hospital stay | perioperatively
  The patient post surgical length of stay in the hospital will be compared between treatment groups.
Absolute value of Interleukin 1 beta (IL-1b) | day 1 after surgery
  Absolute value IL-1b at postoperative day 1 only for participants that have an overnight hospital stay
CD3、CD4、CD4/CD8 and CD16+56 | Preoperative day one，day 1 after surgery
  Postoperative day 1 CD3, CD4, CD4/CD8 and CD16+56 only for participants who were hospitalised overnight and pathologically had lung cancer
Absolute value of Interleukin 6 (IL-6) | day 1 after surgery
  Absolute value IL-6 at postoperative day 1 only for participants that have an overnight hospital stay
C-reactive protein (CRP) | day 1 after surgery
  Absolute value C-reactive protein at postoperative day 1 only for participants that have an overnight hospital stay
Postoperative chest Pain Score | Preoperative day one；Day 1 after surgery; Day 2 after surgery; Day 3 after surgery
  Average postoperative chest pain scores for the first two postoperative days using numerical rating scale (NRS) pain score. Score range from 0 (no pain) to 10 (worst pain possible).
postoperative complications | perioperatively
  Postoperative complications include arrhythmia, bowel obstruction, atrial fibrillation, and other cardiorespiratory systems.
mean arterial pressure | Start of surgery to end of surgery
  Changes in haemodynamics during surgery
systolic blood pressure | Start of surgery to end of surgery
  Changes in haemodynamics during surgery
diastolic blood pressure | Start of surgery to end of surgery
  Changes in haemodynamics during surgery
heart rate | Start of surgery to end of surgery
  Changes in haemodynamics during surgery
liver function | perioperatively
  Transaminases in biochemical indicators
kidney function | perioperatively
  Creatinine in biochemical indicators
Incidence of remedial analgesia | perioperatively
  Remedial analgesia was given when the patient's numerical analogue score (NRS) was greater than 3 in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: QINGhe ZHOU, professor, Principal Investigator — deputy chair of board
Locations (1):
- The First Hospital of Jiaxing, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xie Y, Yan D, Shen J. Video-assisted thoracic surgery versus thoracotomy for treatment of patients with pulmonary sequestration: A systematic review and meta-analysis. Asian J Surg. 2023 Aug;46(8):3387-3388. doi: 10.1016/j.asjsur.2023.03.097. Epub 2023 Mar 25. No abstract available. PMID 36973139
- [Result] Elsharkawy H, Ince I, Pawa A. Rhomboid intercostal and sub-serratus (RISS) plane block for analgesia after lung transplant. J Clin Anesth. 2019 Sep;56:85-87. doi: 10.1016/j.jclinane.2019.01.042. Epub 2019 Jan 28. No abstract available. PMID 30703673
- [Derived] Xie L, Xi Y, He X, An M, Jia X, Li Z, Chen T, Zhou Q. Liposomal Bupivacaine vs. Plain Bupivacaine with Dexamethasone for Rhomboid Intercostal Block in the Management of Postoperative Pain After Video-Assisted Thoracoscopic Surgery: A Randomized Non-inferiority Trial. Pain Ther. 2025 Oct;14(5):1513-1530. doi: 10.1007/s40122-025-00763-1. Epub 2025 Aug 4. PMID 40758210